CLINICAL TRIAL: NCT01794650
Title: The Metabolic and Glycaemic Responses to Changes in the Glycaemic Index of the Meal Consumed After Performing Evening Exercise in Type 1 Diabetes Mellitus
Brief Title: Guidelines for Post-exercise Dietary Intake in T1DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: West-Walker2
Record Dates: First submitted 2013-02-15; First posted 2013-02-20 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: T1DM, Exercise, Hypoglycaemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Meal composition (Other): Changing the glycaemic index of the meals consumed after exercise and before sleep. (High GI - High GI, Low GI - Low GI, High GI - Low GI, Low GI - High GI).
  Interventions: Dietary Supplement: Meal composition

INTERVENTIONS:
Dietary Supplement: Meal composition

SUMMARY:
The investigators hypothesise that manipulating the glycaemic index of the meal after exercise and before sleep will help prevent Type 1 diabetes individuals experiencing hypoglycaemia.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-50 years old (male or female).
* Free from any diabetes related complications (apart from mild background diabetic retinopathy).
* HbA1c <8.5%.
* Not taking any prescribed medication other than insulin, and treated with a stable insulin regimen composed of a combination of slow/long acting insulin (glargine or detemir) and fast-acting insulin analogues (lispro or aspart), for a minimum of 6 months before the start of the study.
* Demonstrate normal cardiac function in response to exercise.

Exclusion Criteria:

* Aged younger than 18, or older than 50 years.
* Suffering from, or diagnosed with a diabetes related complication (apart from mild background diabetic retinopathy).
* HbA1c >8.5%.
* Currently taking prescribed medication, and not currently treated with a stable basal bolus regimen composed of a combination glargine or determir, and lispro or aspart for at least 6 months before the start of the study.
* Failure to demonstrate normal cardiopulmonary responses during exercise, or have a medical condition which could prevent completion of exercise or be exacerbated because of.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2013-03; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
24 hour blood glucose area under the curve | 24 hours
  24 hour, post-exercise, glucose area under the curve.

SECONDARY OUTCOMES:
Ketogenesis | 60 minutes before and 24 hours post-exercise
  Blood beta-hydroxybutyrate concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J West, PhD, BSc, Principal Investigator — Northumbria University
Locations (1):
- Clinical Research Facility, Royal Victoria Infirmary, Newcastle upon Tyne, Tyne and Wear, United Kingdom